CLINICAL TRIAL: NCT02592889
Title: (MitraClip in Non-Responders to Cardiac Resynchronization Therapy)
Acronym: MITRA-CRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, DR. XAVIER FREIXA, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MITRA-CRT
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: MITRAL REGURGITATION
Keywords: MITRAL REGURGITATION
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: mitraclip versus control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL (No Intervention): OPTIMIZED MEDICAL TREATMENT
- DEVICE (Active Comparator): MITRAL VALVE REPAIR WITH THE MITRACLIP SYSTEM + OPTIMIZED MEDICAL TREATMENT
  Interventions: Device: MITRACLIP

INTERVENTIONS:
Device: MITRACLIP — MITRAL VALVE REPAIR WITH THE MITRACLIP SYSTEM
  Arms: DEVICE

SUMMARY:
Functional mitral regurgitation (FMR) is a common finding in patients with dilated cardiomyopathy and reduced left ventricular ejection fraction (LVEF). The presence of a relevant FMR (grade ≥2) is associated with a higher morbidity and mortality. Cardiac resynchronization therapy (CRT) has been shown to be effective in patients with dilated cardiomyopathy and reduced LVEF. In selected patients, CRT has been linked to clinical improvement and reduced mortality. Importantly, 38% of patients with clinical indication for CRT present moderate or severe (FMR). Although FMR might be reduced after CRT, the persistence of a relevant FMR (≥2) after CRT ranges between 40% and 50% and is an independent predictor of no clinical response. In these patients, surgical FMR correction is frequently turned down as a result of a high surgical risk. Percutaneous repair of the mitral valve with the MitraClip system has demonstrated promising results in patients with dilated cardiomyopathy and reduced LVEF5. In a cohort of patients with no response to CRT and FMR ≥2, Auricchio et al showed significant clinical improvement with LVEF recovery and reduction in left ventricle (LV) volumes after MitraClip. The absence of randomization, the retrospective nature of the study and the subsequent selection biases were however major limitations that impeded solid conclusions. The objective of the present study is to assess the efficacy and safety of the MitraClip system in non-responders to CRT and FMR ≥2.

DETAILED DESCRIPTION:
STUDY HYPOTHESIS:

In patients with no response to CRT and significant FMR (grade ≥2, 100%), the MitraClip system will be associated with improved functional class, LVEF recovery and reduced LV volumes. To our knowledge, no registered randomized studies with a similar design are being conducted.

MAIN OBJECTIVE:

To compare the efficacy and safety of optimal medical treatment and MitraClip versus optimal medical treatment alone (control) in non-responders to CRT and symptomatic FMR ≥2.

ELIGIBILITY:
Inclusion Criteria:

1. CRT implanted between 6 months and 5 years before inclusion.
2. Absence of clinical response to CRT defined by baseline NYHA 3 or NYHA 2 with a hospital admission for HF within the last 12 months.
3. Adequate CRT therapy (correct stimulation in >98% heart beats).
4. Correct position of the cardiac leads.
5. Patients with atrial fibrillation will be included but balanced in both groups (the presence of AF is and independent factor of clinical response).
6. Wide QRS (>0.12) and LBBB pre-CRT.
7. LVEF 15-40% (as a surgical risk criteria).
8. Left ventricle end-diastolic diameters <75 mm (as anatomical criteria for MitraClip feasibility).

Exclusion Criteria:

1. Severe Renal Insufficiency (DFGe <30).
2. Life expectancy < 1 year.
3. Anatomical contraindication for MitraClip (in order to avoid selection biases, all patients must be Mitraclip candidates).
4. Hemodynamic instability before inclusion defined by SBP <70 mmHg or the need of inotropic treatment within the previous 3 months.
5. Inadequate treatment compliance or difficult follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants without adverse events related with the therapy and clinical improvement | 1 YEAR CLINICAL
  Number of participants without adverse events related with the therapy (stroke, device embolization, emergent surgery/pericardiocentesis or procedural related mortality) and clinical improvement defined by improvement >10% in 6 min-walking test compared to the baseline situation and no readmissions for heart failure, heart transplantation or mortality.
  SAFETY Definition: Stroke, device embolization, emergent surgery/pericardiocentesis and procedural related mortality.

CONTACTS AND LOCATIONS:
Overall Officials: XAVIER FREIXA, MD, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Freixa X, Tolosana JM, Cepas-Guillen PL, Hernandez-Enriquez M, Sanchis L, Flores-Umanzor E, Farrero M, Andrea R, Roque M, Carretero MJ, Regueiro A, Brugaletta S, Rodes-Cabau J, Mont L, Sitges M, Sabate M, Castel MA. Edge-to-Edge Transcatheter Mitral Valve Repair Versus Optimal Medical Treatment in Nonresponders to Cardiac Resynchronization Therapy: The MITRA-CRT Trial. Circ Heart Fail. 2022 Dec;15(12):e009501. doi: 10.1161/CIRCHEARTFAILURE.121.009501. Epub 2022 Sep 20. No abstract available. PMID 36124767